CLINICAL TRIAL: NCT04011150
Title: Development of Variable Volume Automated Mandatory Boluses (VVAMB) for Patient-controlled Epidural Analgesia During Labour and Delivery
Brief Title: Development of Variable Volume Automated Mandatory Boluses for Patient-controlled Epidural Analgesia During Labour
Acronym: VVAMB
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM/CT001/2018
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Labor Pain; Breakthrough Pain
Keywords: Labor Pain; Breakthrough Pain; Infusion pump
MeSH Terms: conditions — Labor Pain; Breakthrough Pain | interventions — Ropivacaine; Fentanyl; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable volume Automated Mandatory Bolus (VVAMB) (Experimental): The anaesthetic drug and pain medication are prepared in an epidural infusion pump with the VVAMB programme. The programme uses higher doses with lower frequency of medication (ropivacaine and fentanyl), and a patient control button for the patient to control the additional pain relief demands depending on the requirements during labour.
  Interventions: Device: Epidural infusion pump; Drug: Ropivacaine; Drug: Fentanyl
- Automated mandatory bolus (AMB) of variable-frequency (VAMB) (Active Comparator): The anaesthetic drug and pain medication are prepared in an epidural infusion pump with the VAMB programme. The programme uses lower doses with more frequency of medication (ropivacaine and fentanyl), and a patient control button for the patient to control the additional pain relief demands depending on the requirements during labour.
  Interventions: Device: Epidural infusion pump; Drug: Ropivacaine; Drug: Fentanyl

INTERVENTIONS:
Device: Epidural infusion pump — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Other Names: Epidural delivery system
Drug: Ropivacaine — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Other Names: Amide local anaesthetic
Drug: Fentanyl — Epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution.
  Other Names: Opioid

SUMMARY:
A novel epidural delivery regimen was developed: Variable volume automated mandatory bolus (AMB) (VVAMB) will advance individualisation of labour epidural analgesia, by which a larger volume of bolus may contribute to better spread of the local anaesthetics within brief period and thereby reduces the chances of motor blockade that could reduce instrumental deliveries.

DETAILED DESCRIPTION:
Epidural analgesia is the gold standard of pain relief for labour pain. Despite this, up to 50% of parturients continue to experience pain leading to suffering and increased caregiver workload. There is also higher risk of motor blockade found in those receiving epidural analgesia, and these factors is associated with dysfunctional labour requiring obstetric intervention (instrumental delivery). Automated mandatory bolus (AMB) of variable-frequency (VAMB) has been shown to provide better pain relief as compared with conventional patient-controlled epidural analgesia (PCEA) with basal infusion, however its long lockout time per hour is associated with unsuccessful patient bolus requests, with similar motor block to conventional regimens.

The investigators therefore proposes to develop a novel epidural delivery regimen: Variable volume AMB (VVAMB) will advance individualisation of labour epidural analgesia, by which a larger volume of bolus may contribute to better spread of the local anaesthetics within brief period and thereby reduces the chances of motor blockade that could reduce instrumental deliveries. This algorithm development including pilot and clinical trial will compare VVAMB with VAMB regimens, in reducing the incidence of motor block in 216 term women requesting for labour epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (American Society of Anesthesiologists (ASA) physical status 1 and 2) primiparous parturient at term (≥36 weeks gestation);
* Singleton fetus;
* In early labor stage (cervical dilation ≤5cm);
* Request labor epidural analgesia and able to administer combined spinal epidural analgesia (CSEA) according to protocol.

Exclusion Criteria:

* Non-cephalic fetal presentation;
* Obstetric (e.g. pre-eclampsia, premature rupture of amniotic membranes for more than 48 hours, gestational diabetes on insulin, pregnancy-induced hypertension on medication) and uncontrolled medical (e.g. cardiac disease) complications;
* Have contraindications to neuraxial blockade or have received parenteral opioids within last 2 hours;
* Dural puncture/ suspected dural puncture at initiation of CSEA.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females having natural delivery in KKH will be recruited.
Enrollment: 216 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of motor block in each group | During labour (1 day)
  The number of event of motor block throughout the labour. Previous studies have shown that epidural analgesia using high concentrations of local anaesthetics could lead to decreased motor functions, and are subsequently associated with an increased incidence of instrumented delivery and longer second stage of labour. In this study, the intensity of motor block is assessed by the patient's ability to move their lower extremities via a modified Bromage scale. In the modified version, a scoring of 0 implies no motor block (Free movement of both legs and feet), scoring of 1 implies partial block (Just able to flex knees with free movement of feet), 2 implies almost complete block (Unable to flex knees but with free movement of feet) and 3 implies a full block (Unable to move legs/ feet).

SECONDARY OUTCOMES:
Number of subjects with Instrumental delivery | During labour (1 day)
  The number of subjects in each group having instrumental delivery (forceps, vacuum delivery)
Number of subjects with Breakthrough pain | During labour (1 day)
  The number of subjects in each group having unscheduled epidural supplementation by anaesthetist due to labor pain
APGAR score | After delivery (1 day)
  The Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) score is a test given to newborns soon after birth. In the test, five are being evaluated: Appearance (skin color), Pulse (heart rate), Grimace response (reflexes), Activity (muscle tone) and Respiration (breathing rate and effort). Each is scored on a scale of 0 to 2, with 2 being the best score; a total score of ten represents the best possible condition.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ling Leong, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No